CLINICAL TRIAL: NCT05747885
Title: The Rehabilitation Complexity Scale (RCS) in Pulmonary Rehabilitation: Utility and Limitations
Brief Title: Application of RCS in Pulmonary Rehabilitation
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Other Study IDs: ICS Maugeri CE 2713
Record Dates: First submitted 2023-01-31; First posted 2023-02-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Respiratory Disease
Keywords: Appropriateness; motor pulmonary rehabilitation; Rehabilitation Complexity Scale
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In August 2021, the Italian Ministry of Health published the Ministerial Decree to define the "Criteria for the appropriateness concerning the access to hospital rehabilitation admission" (in neurological, respiratory, cardiological, and orthopedic Units), classifying patients by complexity, the severity of disability and the number of ICD-9 discharge codes. The Appropriateness Decree adopted some fundamental criteria used in the United Kingdom for over 10 years (2009) where the Ministry of Health defined 3 levels of specialized rehabilitation based on the different complexity of the patient's needs. Among the scales, the Rehabilitation Complexity Scale (RCS) has been proposed by the British Society of Rehabilitation Medicine (BSRM), clearly oriented to patients with motor disabilities (neurological and orthopedic), of which the RCS-E (i.e. Extended version) is the more up to date.

The Italian Ministry of Health has proposed the application of the RCS scale as a tool for measuring rehabilitation complexity based on the intensity and level of skills required in terms of nursing, medical and therapeutic care.

In this Clinical Study the Investigators intend to 1. test the application of the new RCS scale to rehabilitation admissions in 16 Italian Pulmonary Rehabilitation Units 2. correlate this scale to the most universally used clinical and functional measures evaluated in the respiratory field 3. investigate the responsiveness of the RCS scale at the end of rehabilitation 4. promote an audit to revise the clinical and rehabilitation conditions -described by items of the RCS-E- to get a specific RCS referable to respiratory patients with MDC4.

DETAILED DESCRIPTION:
Background In August 2021, the Italian Ministry of Health published the Ministerial Decree to define the "Criteria for the appropriateness concerning the access to hospital rehabilitation admission" (in neurological, respiratory, cardiologic, and orthopedic Units), classifying patients by complexity, the severity of disability and the number of ICD-9 discharge codes. The Appropriateness Decree adopts some fundamental criteria used in the United Kingdom for over 10 years (2009) where the Ministry of Health has defined 3 levels of specialized rehabilitation based on the different complexity of the patient's needs. Among the possible scales, the Rehabilitation Complexity Scale (RCS) has been proposed by the British Society of Rehabilitation Medicine (BSRM), clearly oriented to patients with motor disabilities (neurological and orthopedic), of which the RCS-E (i.e. Extended version) is the more up to date.

The Italian Ministry of Health has recently proposed the application of the RCS scale as a tool for measuring rehabilitation complexity based on the intensity and level of skills required in terms of nursing, medical and therapeutic care.

In this Clinical Study the Investigators intend to 1. test the application of the new RCS scale to rehabilitation admissions in 16 Italian Pulmonary Rehabilitation Units 2. correlate this scale to the most universally used clinical and functional measures evaluated in the respiratory field 3. investigate the responsiveness of the RCS scale at the end of rehabilitation 4. promote an audit to revise the clinical and rehabilitation conditions -described by items of the RCS-E- to obtain a specific RCS referable to respiratory patients with MDC4.

Methods This is a multicenter observational study. Patients hospitalized in 16 Pulmonary Rehabilitation Units for a period of respiratory rehabilitation, as defined by the latest guidelines of the American Thoracic Society / European Respiratory Society (ATS/ERS), will be considered. Clinical data [Diagnosis at admission, Demographic and anthropometric data, Provenience (home or hospital), Days of hospitalization in the rehabilitation unit], other than tests/evaluations/scales usually administered at the admission and discharge of the rehabilitation process will be collected.

All information will be used to fill in the RCS-E both at admission and discharge.

The Outcome measures are reported in the dedicated section.

The Sample size has been estimated at 400 patients (considering 25 patients with any DRG/center admitted on 2 specific days at each institute).

Summary statistics will be presented as a descriptive analysis of the mean and standard deviation or median and quartiles for continuous variables and as counts with percentages for categorical or dichotomous variables. Patients will be stratified according to the 3 main DRGs (invasive ventilation 566/565, 88 CRF, 87 COPD) and comparisons will be performed by ANOVA test for continuous variables and chi-square test for categorical or dichotomous variables.

Testing for significant differences in the distributions of discrete variables will be performed with the Chi-Square Test and the Student t-Test will be used for the comparison of pre to post-continuous variables (difference between Baseline and Post program).

Correlations between RCS-E and the standard respiratory/disability scales [Barthel Dyspnea Index, Medical Resource Council (MRC), COPD Assessment Test (CAT), and meters covered in the 6 minutes] will be performed by Spearman's test. An inadequate/adequate correlation with respect to the usual measurements will make it possible to define the "applicability/goodness"" of the scale proposed by the Ministry.

For all tests, a p-value <.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* all patients hospitalized for Pulmonary Rehabilitation in two dedicated days (core drilling day 1 = 30 January 2023 and core drilling day 2 = 28 February 2023)

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in 16 Pulmonary Rehabilitation Units will be considered. These patients will participate in a pulmonary rehabilitation program, as defined by the latest guidelines of the American Thoracic Society / European Respiratory Society (ATS/ERS).
Sampling Method: Non-Probability Sample
Enrollment: 547 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Rehabilitation Complexity Scale (RCS)-E description | At the date of admission in rehabilitation
  To evaluate the level of complexity and care needs with the RCS-E scale in patients hospitalized attending pulmonary rehabilitation centers. The Rehabilitation Complexity Scale (RCS) describes the level of support the patient needs for either basic self-care or to maintain their safety. 0=best outcome; 22= worst outcome.
RCS-E correlation with Baseline Barthel Dyspnea Index | At the date of admission in rehabilitation
  To correlate RCS-E with one of the most universally used indicators at admission in the respiratory field for symptoms (Barthel Dyspnea Index)
RCS-E correlation with Baseline Medical Research Council (MRC) | At the date of admission in rehabilitation
  To correlate RCS-E with one of the most universally used indicators at admission in the respiratory field for symptoms (MRC)
RCS-E correlation with Baseline COPD Assessment Test (CAT) | At the date of admission in rehabilitation
  To correlate RCS-E with one of the most universally used indicators at admission in the respiratory field for the quality of life (CAT)
RCS-E correlation with Baseline six minutes walking test (6MWT) distance | At the date of admission in rehabilitation
  To correlate RCS-E with one of the most universally used indicators at admission in the respiratory field for the effort tolerance (6MWT distance)
RCS-E correlation with clinical outcome (discharged home, transferred or dead) | From the date of admission in rehabilitation to the date of discharge (up to three weeks)
  To correlate RCS-E with one of the most universally used indicators in the respiratory field for clinical outcome (discharged home, transferred or dead)
Change in RCS-E | From the date of admission in rehabilitation to the date of discharge (up to three weeks)
  To evaluate the responsivity of RCS-E to Pulmonary rehabilitation in terms of the significative difference between baseline and end of program.The Rehabilitation Complexity Scale (RCS) describes the level of support the patient needs for either basic self-care or to maintain their safety. 0=best outcome; 22= worst outcome.

SECONDARY OUTCOMES:
Comparison of RCS-E among groups | At the date of admission in rehabilitation
  To describe the distribution of RCS-E as a function of the 3 main DRGs (ventilated trachea 566/565, CRF, COPD)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Vitacca, MD, Study Director — ICS Maugeri IRCCS, respiratory rehabilitation of the Institute of Lumezzane; Paolo Banfi, MD, Study Director — Fondazione Don Carlo Gnocchi ONLUS, IRCCS Centro S. Maria Nascente, Respiratory rehabilitation
Locations (16):
- Italy (16):
  - ICS Maugeri IRCCS, Respiratory rehabilitation of the Institute of Telese, Telese Terme, Benevento
  - ICS Maugeri IRCCS, Respiratory rehabilitation of the Institute of Lumezzane, Lumezzane, Brescia
  - Fondazione Don Carlo Gnocchi ONLUS, Centro "Spalenza", Respiratory rehabilitation, Rovato, Brescia
  - Ospedale "Santa Marta" di Rivolta d'Adda, Respiratory rehabilitation, Rivolta d'Adda, Cremona
  - Istituto nazionale Riposo e Cura per Anziani di Casatenovo, Respiratory rehabilitation, Casatenovo, Lecco
  - Ospedale di Codogno- Centro di riabilitazione cardio-respiratorio, Codogno, Lodi
  - Presidio Ospedaliero di Sant'Angelo Lodigiano, Respiratory rehabilitation, Sant'Angelo Lodigiano, Lodi
  - Ospedale Villa Pineta, Respiratory rehabilitation, Pavullo nel Frignano, Modena
  - ICS Maugeri IRCCS, Respiratory rehabilitation of the Institute of Veruno, Veruno, Novara
  - ICS Maugeri IRCCS, Respiratory rehabilitation of the Institute of Montescano, Montescano, Pavia
  - ICS Maugeri IRCCS, Respiratory rehabilitation of the Institute of Tradate, Tradate, Varese
  - ICS Maugeri IRCCS, Respiratory rehabilitation of the Institute of Bari, Bari
  - Fondazione Don Carlo Gnocchi ONLUS, IRCCS "Don Carlo Gnocchi", Respiratory rehabilitation, Florence
  - Fondazione Don Carlo Gnocchi ONLUS, IRCCS Centro S. Maria Nascente, Respiratory rehabilitation, Milan
  - Ospedale Monaldi, Aziende Ospedaliera Specialistica dei Colli, Respiratory rehabilitation, Napoli
  - ICS Maugeri IRCCS, Respiratory rehabilitation of the Institute of Pavia, Pavia

REFERENCES:
- [Background] Turner-Stokes L, Disler R, Williams H. The Rehabilitation Complexity Scale: a simple, practical tool to identify 'complex specialised' services in neurological rehabilitation. Clin Med (Lond). 2007 Dec;7(6):593-9. doi: 10.7861/clinmedicine.7-6-593. PMID 18193708
- [Background] Turner-Stokes L, Williams H, Siegert RJ. The Rehabilitation Complexity Scale version 2: a clinimetric evaluation in patients with severe complex neurodisability. J Neurol Neurosurg Psychiatry. 2010 Feb;81(2):146-53. doi: 10.1136/jnnp.2009.173716. Epub 2009 Jul 8. PMID 19587391
- [Background] Turner-Stokes L, Scott H, Williams H, Siegert R. The Rehabilitation Complexity Scale--extended version: detection of patients with highly complex needs. Disabil Rehabil. 2012;34(9):715-20. doi: 10.3109/09638288.2011.615880. Epub 2011 Nov 24. PMID 22115200
- [Background] Pedersen AR, Nielsen JF, Jensen J, Maribo T. Referral decision support in patients with subacute brain injury: evaluation of the Rehabilitation Complexity Scale - Extended. Disabil Rehabil. 2017 Jun;39(12):1221-1227. doi: 10.1080/09638288.2016.1189610. Epub 2016 Jul 6. PMID 27384499
- [Background] Turner-Stokes L, Sutch S, Dredge R, Eagar K. International casemix and funding models: lessons for rehabilitation. Clin Rehabil. 2012 Mar;26(3):195-208. doi: 10.1177/0269215511417468. Epub 2011 Nov 9. PMID 22070989
- [Background] Koh GC, Chen CH, Petrella R, Thind A. Rehabilitation impact indices and their independent predictors: a systematic review. BMJ Open. 2013 Sep 24;3(9):e003483. doi: 10.1136/bmjopen-2013-003483. PMID 24068767
- [Background] Roda F, Agosti M, Corradini E, Lombardi F, Maini M, Brianti R. Cross-cultural adaptation and preliminary test-retest reliability of the Italian version of the Complexity Rehabilitation Scale-Extended (13th version). Eur J Phys Rehabil Med. 2015 Aug;51(4):439-46. Epub 2014 Mar 4. PMID 24621987
- [Background] Galletti L, Benedetti MG, Maselli S, Zanoli G, Pignotti E, Iovine R. Rehabilitation Complexity Scale: Italian translation and transcultural validation. Disabil Rehabil. 2016;38(1):87-96. doi: 10.3109/09638288.2015.1024340. Epub 2015 Apr 15. PMID 25875050
- [Background] Roda F, Agosti M, Merlo A, Maini M, Lombardi F, Tedeschi C, Benedetti MG, Basaglia N, Contini M, Nicolotti D, Brianti R; GRECo. Psychometric validation of the Italian Rehabilitation Complexity Scale-Extended version 13. PLoS One. 2017 Oct 18;12(10):e0178453. doi: 10.1371/journal.pone.0178453. eCollection 2017. PMID 29045409
- [Background] Chang EY, Chang EH, Cragg S, Cramer SC. Predictors of Gains During Inpatient Rehabilitation in Patients with Stroke- A Review. Crit Rev Phys Rehabil Med. 2013;25(3-4):203-221. doi: 10.1615/CritRevPhysRehabilMed.2013008120. PMID 25541570
- [Background] Kwon S, Hartzema AG, Duncan PW, Min-Lai S. Disability measures in stroke: relationship among the Barthel Index, the Functional Independence Measure, and the Modified Rankin Scale. Stroke. 2004 Apr;35(4):918-23. doi: 10.1161/01.STR.0000119385.56094.32. Epub 2004 Feb 19. PMID 14976324
- [Background] Balasch i Bernat M, Balasch i Parisi S, Sebastian EN, Moscardo LD, Ferri Campos J, Lopez Bueno L. Determining cut-off points in functional assessment scales in stroke. NeuroRehabilitation. 2015;37(2):165-72. doi: 10.3233/NRE-151249. PMID 26484508
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Paneroni M, Simonelli C, Vitacca M, Ambrosino N. Aerobic Exercise Training in Very Severe Chronic Obstructive Pulmonary Disease: A Systematic Review and Meta-Analysis. Am J Phys Med Rehabil. 2017 Aug;96(8):541-548. doi: 10.1097/PHM.0000000000000667. PMID 28099192
- [Background] Holland AE, Cox NS, Houchen-Wolloff L, Rochester CL, Garvey C, ZuWallack R, Nici L, Limberg T, Lareau SC, Yawn BP, Galwicki M, Troosters T, Steiner M, Casaburi R, Clini E, Goldstein RS, Singh SJ. Defining Modern Pulmonary Rehabilitation. An Official American Thoracic Society Workshop Report. Ann Am Thorac Soc. 2021 May;18(5):e12-e29. doi: 10.1513/AnnalsATS.202102-146ST. PMID 33929307
- See also: King's College London - RCS-E - Rehabilitation Complexity Scale Extended — https://www.kcl.ac.uk/cicelysaunders/resources/tools/RCS-Ee
- See also: Report of Global Initiative for Lung Disease (GOLD) criteria for COPD — https://goldcopd.org/2022-gold-reports